CLINICAL TRIAL: NCT05438888
Title: Safety and Effectiveness of Apixaban in Very Elderly Patients With NVAF Compared to Warfarin Using Administrative Claims Data
Brief Title: Safety and Effectiveness of Apixaban in Very Elderly Patients With Non-valvular Atrial Fibrillation (NVAF) Compared to Warfarin Using Administrative Claims Data
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661181
Record Dates: First submitted 2022-06-25; First posted 2022-06-30 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2023-10

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Stroke; Apixaban; Warfarin
MeSH Terms: conditions — Stroke | interventions — Warfarin; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Warfarin cohort (Reference): Patients with NVAF treated with warfarin
  Interventions: Drug: Warfarin
- Apixaban cohort: Patients with NVAF treated with apixaban
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Warfarin — This is observational study and the patients in the warfarin cohort include those who are exposed to warfarin in the real world settings.
  Groups: Warfarin cohort (Reference)
Drug: Apixaban — This is observational study and the patients in the apixaban cohort include those who are exposed to apixaban in the real world settings.
  Groups: Apixaban cohort

SUMMARY:
The objective of this study is to investigate safety and effectiveness of apixaban compared to warfarin in very elderly patients with Non-valvular atrial fibrillation (NVAF). In addition to the absolute age, effects on higher age-related risk factors on relative risk of apixaban to warfarin is also investigated through subgroup analyses.

DETAILED DESCRIPTION:
This is a retrospective non-intervention observational study to evaluate the difference in safety and effectiveness between apixaban and warfarin using a database provided by Medical Data Vision Co. Ltd. (MDV Co. Ltd.). Eligible patients will be extracted from the database and allocated to the pre-defined cohorts based on the actual age, age of NVAF diagnosis and types of anticoagulant therapy.

Patient characteristics will be balanced by an Inverse probability of treatment weighting (IPTW) method, and risk of stroke/SE (primary effectiveness endpoint) and major bleeding (primary safety endpoint) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following inclusion criteria to be eligible for inclusion in the study.

  1. Diagnosed with Atrial fibrillation (AF) anytime in the baseline period or on the index date, also have definitive diagnosis of AF anytime in the baseline period, on the index date, or post-index period.
  2. Prescribed apixaban or warfarin on or after the day of AF diagnosis. The first observed prescription will be used to identify the patient's index date and treatment cohort
  3. No use of the any Oral anticoagulants (OAC)s during the baseline period (the 180 days before the index date)
  4. Age of 18 years or older on the index date.
  5. Index date is at age 80 or older

Exclusion Criteria:

* Patients meeting any of the following criteria will not be included in the study:

  1. Having a diagnosis of valvular atrial fibrillation, post-operative atrial fibrillation, rheumatic atrial fibrillation or mechanical-valvular atrial fibrillation during the baseline and post-index period
  2. Having a cardiac surgery procedure record during the baseline period
  3. Having a joint replacement procedure record during the baseline period
  4. Having a procedure of prosthetic heart valve during the baseline period
  5. Having a diagnosis of venous thromboembolism during the baseline period
  6. Female patients with pregnancy during the follow-up period
  7. Patients prescribed "off-label" doses of OACs (per Japanese package insert of each OAC) or patients treated with OAC but in "off-label" or "contraindicated" manners.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 80 years or older who are newly diagnosed with non-valvular atrial fibrillation (NVAF) and initiate anticoagulation therapy with warfarin or apixaban.
Sampling Method: Probability Sample
Enrollment: 77814 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Matsuo-Ohsawa A, Katada J, Kohsaka S. Safety and Effectiveness of Apixaban in Very Elderly Patients with Atrial Fibrillation: A Retrospective Analysis of Japanese Administrative Claims Data. Cardiol Ther. 2025 Dec;14(4):565-581. doi: 10.1007/s40119-025-00420-w. Epub 2025 Jul 8. PMID 40627071
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants who received apixaban or warfarin (80 years or older) after getting diagnosed with non-valvular atrial fibrillation (NVAF) were observed in this retrospective observational study.
Pre-assignment Details: Data of eligible participants were extracted from Medical Data Vision Company Limited (MDV Co. Ltd.) database for duration of 26-Feb-2013 to 31-Dec-2021. Extracted data was evaluated for objectives of this study in approximately 3.5 months of this study.
Groups:
- Warfarin Cohort: Participants included in this cohort were those who received warfarin in real world practice after getting diagnosed with NVAF. Data of the participants included were retrieved from MDV database and was observed retrospectively in this study.
- Apixaban Cohort: Participants included in this cohort were those who received apixaban in real world practice after getting diagnosed with NVAF. Data of the participants included were retrieved from MDV database and was observed retrospectively in this study.
Period: Overall Study
Arm/Group | Warfarin Cohort | Apixaban Cohort
Started | 39936 | 37878
Completed | 39936 | 37878
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants whose data were extracted from database and observed in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin Cohort | Apixaban Cohort | Total
Number analyzed (Participants) | 39936 | 37878 | 77814
Age, Continuous [Mean (Standard Deviation); unit: Years] | 85.3 (4.15) | 85.7 (4.22) | 85.5 (4.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18804 | 19171 | 37975
  Male | 21132 | 18707 | 39839
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate (Per 1,000 Participant-Year) of Composite of Stroke and Systemic Embolism (SE): Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of composite stroke and SE events after index date was reported. Stroke events included ischemic and hemorrhagic stroke. International Classification of Diseases 10th Revision (ICD-10) diagnosis code was used to label the events. Index date was defined as a date when participants initiated warfarin or apixaban. Follow-up period: the next day of the index date till occurrence of target outcome, discontinuation of the warfarin or apixaban, switching from the warfarin or apixaban, withdrawal from the database, whichever observed first.
Time Frame: Follow-up period during data observation period from 26-Feb-2013 to 31-Dec-2021 (approximately 8 years 10 months); extracted data evaluated in approximately 3.5 months of this study
Population: Eligible participants registered on MDV database, whose data was observed in the study. Analysis was performed using inverse probability treatment weighting with stabilized weights (s-IPTW) method to balance participant characteristics among reporting groups. Here, "Overall Number of Participants Analyzed" is the number of participants after application of s-IPTW method to raw numbers and is different from the actual participants included in the reporting arm.
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Groups:
- Warfarin: Balanced Cohort: Participants included in this cohort were those who received warfarin in real world practice after getting diagnosed with NVAF. Data of the participants included were retrieved from MDV database and was observed retrospectively in this study. S-IPTW method was applied to balance the participant's characteristics.
- Apixaban: Balanced Cohort: Participants included in this cohort were those who received apixaban in real world practice after getting diagnosed with NVAF. Data of the participants included were retrieved from MDV database and was observed retrospectively in this study. S-IPTW method was applied to balance the participant's characteristics.
Arm/Group | Warfarin: Balanced Cohort | Apixaban: Balanced Cohort
Number analyzed (Participants) | 43671 | 33834
Events Per 1000 Participant-Years | 75.227 [72.579 to 77.972] | 55.801 [53.328 to 58.388]
Statistical Analysis 1: Comparison: Warfarin: Balanced Cohort vs Apixaban: Balanced Cohort; Test type: Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.753, 95% CI 2-sided [0.711 to 0.798]

2. Primary Outcome: Incidence Rate (Per 1,000 Participant-Year) of Major Bleeding: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of major bleeding event after index date was reported. Major bleeding was defined as any bleeding that required hospitalization for treatment. ICD-10 diagnosis code was used to label the events. Index date was defined as a date when participants initiated warfarin or apixaban. Follow-up period: the next day of the index date till occurrence of target outcome, discontinuation of the warfarin or apixaban, switching from the warfarin or apixaban, withdrawal from the database, whichever observed first.
Time Frame: as for outcome 1
Population: Eligible participants registered on MDV database, whose data was observed in the study. Analysis was performed using s-IPTW method to balance participant characteristics among reporting groups. Here, "Overall Number of Participants Analyzed" is the number of participants after application of s-IPTW method to raw numbers and is different from the actual participants included in the reporting arm.
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Warfarin: Balanced Cohort | Apixaban: Balanced Cohort
Number analyzed (Participants) | 43671 | 33834
Events Per 1000 Participant-Years | 25.328 [23.836 to 26.914] | 17.306 [15.973 to 18.751]
Statistical Analysis 1: Comparison: Warfarin: Balanced Cohort vs Apixaban: Balanced Cohort; Test type: Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.687, 95% CI 2-sided [0.622 to 0.760]

3. Secondary Outcome: Incidence Rate (Per 1,000 Participant-Year) of Cardiogenic Cerebral Embolism: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of cardiogenic cerebral embolism events after index date was reported. ICD-10 diagnosis code was used to label the events. Index date was defined as a date when participants initiated warfarin or apixaban. Follow-up period: the next day of the index date till occurrence of target outcome, discontinuation of the warfarin or apixaban, switching from warfarin or apixaban, withdrawal from the database, whichever observed first.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Warfarin: Balanced Cohort | Apixaban: Balanced Cohort
Number analyzed (Participants) | 43671 | 33834
Events Per 1000 Participant-Years | 21.386 [20.024 to 22.841] | 13.473 [12.306 to 14.751]
Statistical Analysis 1: Comparison: Warfarin: Balanced Cohort vs Apixaban: Balanced Cohort; Test type: Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.638, 95% CI 2-sided [0.570 to 0.714]

4. Secondary Outcome: Incidence Rate (Per 1,000 Participant-Year) of Ischemic Stroke (Cerebral Infarction): Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of ischemic stroke event after index date was reported. ICD-10 diagnosis code was used to label the events. Index date was defined as a date when participants initiated warfarin or apixaban. Follow-up period: the next day of the index date till occurrence of target outcome, discontinuation of the warfarin or apixaban, switching from warfarin or apixaban, withdrawal from the database, whichever observed first.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Warfarin: Balanced Cohort | Apixaban: Balanced Cohort
Number analyzed (Participants) | 43671 | 33834
Events Per 1000 Participant-Years | 39.607 [37.713 to 41.596] | 33.279 [31.395 to 35.277]
Statistical Analysis 1: Comparison: Warfarin: Balanced Cohort vs Apixaban: Balanced Cohort; Test type: Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.854, 95% CI 2-sided [0.791 to 0.922]

5. Secondary Outcome: Incidence Rate (Per 1,000 Participant-Year) of Intracranial Hemorrhage: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of intracranial hemorrhage event after index date was reported. ICD-10 diagnosis code was used to label the events. Index date was defined as a date when participants initiated warfarin or apixaban. Follow-up period: the next day of the index date till occurrence of target outcome, discontinuation of the warfarin or apixaban, switching from warfarin or apixaban, withdrawal from the database, whichever observed first.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Warfarin: Balanced Cohort | Apixaban: Balanced Cohort
Number analyzed (Participants) | 43671 | 33834
Events Per 1000 Participant-Years | 20.787 [19.443 to 22.223] | 13.138 [11.988 to 14.399]
Statistical Analysis 1: Comparison: Warfarin: Balanced Cohort vs Apixaban: Balanced Cohort; Test type: Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.638, 95% CI 2-sided [0.570 to 0.715]

6. Secondary Outcome: Incidence Rate (Per 1,000 Participant-Year) of Gastrointestinal Bleeding: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of major GI bleeding event after index date was reported. ICD-10 diagnosis code was used to label the events. Index date was defined as a date when participants initiated warfarin or apixaban. Follow-up period: the next day of the index date till occurrence of target outcome, discontinuation of the warfarin or apixaban, switching from warfarin or apixaban, withdrawal from the database, whichever observed first.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Warfarin: Balanced Cohort | Apixaban: Balanced Cohort
Number analyzed (Participants) | 43671 | 33834
Events Per 1000 Participant-Years | 42.641 [40.673 to 44.704] | 36.595 [34.610 to 38.695]
Statistical Analysis 1: Comparison: Warfarin: Balanced Cohort vs Apixaban: Balanced Cohort; Test type: Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.868, 95% CI 2-sided [0.807 to 0.934]

7. Secondary Outcome: Incidence Rate (Per 1,000 Participant-Year) of Intraocular Bleeding: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of intraocular bleeding event after index date was reported. ICD-10 diagnosis code was used to label the events. Index date was defined as a date when participants initiated warfarin or apixaban. Follow-up period: the next day of the index date till occurrence of target outcome, discontinuation of the warfarin or apixaban, switching from warfarin or apixaban, withdrawal from the database, whichever observed first.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Warfarin: Balanced Cohort | Apixaban: Balanced Cohort
Number analyzed (Participants) | 43671 | 33834
Events Per 1000 Participant-Years | 4.224 [3.643 to 4.897] | 2.682 [2.190 to 3.284]
Statistical Analysis 1: Comparison: Warfarin: Balanced Cohort vs Apixaban: Balanced Cohort; Test type: Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.646, 95% CI 2-sided [0.503 to 0.830]

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not planned to be collected during the study.
Description: This study involved data that existed as structured data by the time of study start. In these data sources, individual participant data was not retrieved or validated, and it was not possible to link (i.e., identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met.
Arm/Group | Warfarin Cohort | Apixaban Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT05438888/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT05438888/SAP_001.pdf